CLINICAL TRIAL: NCT00202098
Title: Effects of Variable Ventilation on Respiratory System of ARDS Patients
Brief Title: Effects of Variable Ventilation on Respiratory System of Acute Respiratory Distress Syndrome (ARDS) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 11
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: ARDS
Keywords: ARDS; mechanical ventilation; variable ventilation; chaotic ventilation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): ALI/ARDS patients
  Interventions: Procedure: Variable ventilation

INTERVENTIONS:
Procedure: Variable ventilation — Patients will be mechanically ventilated with Variable Ventilation (3 step with increased level of variability) and "traditional" CMV, for a total of 4 step. Each step lasts in 60 minutes. During this period the investigators will record the gas exchange parameters and the mechanics of the respiratory system.

SUMMARY:
The purpose of this study is to determine the effects of variable ventilation on respiratory system of patients affected by acute respiratory distress syndrome.

DETAILED DESCRIPTION:
In this interventional study we want to evaluate the effect of Variable ventilation (1) in patients with ARDS. Patients will be mechanically ventilated with Variable Ventilation (3 step with increased level of variability) and "traditional" CMV, for a total of 4 step. Each step lasts in 60 minutes. During this period we will record the gas exchange parameters and the mechanics of the respiratory system.

1. Arold S, Mora R, Lutchen K, et al. Variable ventilation improves lung mechanics and gas exchange in a rodent model of acute lung injury. Am J Resp Crit Care Med 2000; 165: 366-71.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ARDS criteria

Exclusion Criteria:

* Age less than 18 years
* Severe haemodynamic instability
* Patients with clinical or instrumental evidence of flow-limitation (i.e., PEEPi)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2005-03; Primary Completion 2013-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Gas exchange and respiratory mechanics | within the first 60 minutes from the ventilatory change

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Taccone, MD, Principal Investigator — Policlinico Hospital Milan
Locations (1):
- Policlinico Hospital, Milan, Italy